CLINICAL TRIAL: NCT06992544
Title: Trial of Pistachio Consumption on Cognition, Cardiometabolic Risk Factors, and Life Satisfaction in Older Adults
Brief Title: Trial of Pistachio Consumption in Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: American Pistachio Growers (Other); Boston Children's Hospital, Boston, MA, USA (Other); University of Illinois at Urbana-Champaign (Other); Quest Diagnostics-Nichols Insitute (Industry)
Responsible Party: Principal Investigator, Howard D. Sesso, ScD, MPH, Associate Epidemiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024P002479
Record Dates: First submitted 2025-04-29; First posted 2025-05-28 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cognition; Cardiometabolic Risk Factors; Life Satisfaction
Keywords: Pistachio; Cognition; Life satisfaction; Older adults; Cardiometabolic risk factors; Blood pressure; Biomarkers; Memory; Diet; Nut intake
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Masking Description: Outcome assessments will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pistachio-enriched diet (Active Comparator): 1 packet/day of approximately 1.25 oz (35 g) of dry roasted, unsalted, shelled pistachio kernels
  Interventions: Other: Pistachio-enriched diet
- Usual diet (Other): Usual diet (while abstaining from pistachio consumption and limiting other nut consumption to ≤1 serving/week)
  Interventions: Other: Usual diet

INTERVENTIONS:
Other: Pistachio-enriched diet — 1 packet/day of approximately 1.25 oz (35 g) of dry roasted, unsalted, shelled pistachio kernels
  Arms: Pistachio-enriched diet
Other: Usual diet — Usual diet (while abstaining from pistachio consumption and limiting other nut consumption to ≤1 serving/week)
  Arms: Usual diet

SUMMARY:
The goal of this study is to evaluate whether a pistachio-enriched diet leads to changes in cognitive function, cardiometabolic risk factors, and life satisfaction in older adults over a 6-month period.

DETAILED DESCRIPTION:
In this remote-based, parallel-arm RCT, the investigators will recruit participants from the recently completed COcoa Supplement and Multivitamin Outcomes Study (COSMOS) trial cohort. Eligible COSMOS participants will be invited to participate in the proposed RCT, screened to verify eligibility and willingness to participate, and asked to provide informed consent. Eligible and willing participants will be enrolled and randomized on a rolling basis. Risk factors and Outcome assessments will be conducted at baseline, 3 months and 6 months via the MyCap Mobile Toolbox application, REDCap questionnaires (for life satisfaction, dietary, and other phenotypic assessments), or at a local Quest Diagnostics (for biospecimen collection and return to our biorepository).

ELIGIBILITY:
Inclusion Criteria:

1. Active participant in COSMOS
2. Current age 65 to 80 years
3. Does not reside in the states of Arizona, Hawaii, or Wyoming (since Quest Diagnostics does not have locations in these states)

Exclusion Criteria:

1. Tree nut allergy
2. Current intake of pistachios, peanuts, walnuts, or other nuts >1 serving/week
3. Diagnosis of Alzheimer's disease or any other type of dementia
4. Diagnosis of cancer or CVD (MI, stroke, CABG, PTCA, or stent) within last 12 months
5. Changes in the dose or number of anti-hypertensive, lipid-lowering, or diabetic medications over the past 3 months prior to randomization
6. Does not own a smartphone or tablet
7. Unable or unwilling to abstain from pistachio intake for 6 months
8. Unable or unwilling to limit nut consumption to ≤1 serving/week for 6 months
9. Unable or unwilling to complete online questionnaires and cognitive assessments
10. Unable or unwilling to travel to a local Quest site for biospecimen collection
11. Unable or unwilling to provide consent to participate in the trial
12. Failure to complete the baseline Life Satisfaction Questionnaire
13. Failure to complete the baseline cognitive assessments
14. Failure to complete the baseline biospecimen collection

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 97 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mobile Toolbox | Baseline and 6 months
  The investigators will assess 6-month changes in the Mobile Toolbox total score as a measure of global cognitive function. The total score considers the following individual cognitive domains (tests): associative memory (Face and Names), executive function (Arrow Matching for inhibitory control, Shape-Color Sorting for cognitive flexibility), episodic memory (Arranging Pictures), working memory (Sequences), and processing speed (Number-Symbol Match). A total score is calculated by adding together each individual test score, for a total of 232 possible points. Scores may range from 0-232, in which a higher score indicates better cognitive function.

SECONDARY OUTCOMES:
Blood pressure | Baseline and 6 months
  The investigators will assess 6-month changes in seated systolic and diastolic blood pressure (in mmHg).
Life Satisfaction for the Third Age-Short Form | Baseline and 6 months
  The investigators will assess 6-month changes in total score for the "Life Satisfaction for the Third Age-Short Form" questionnaire, a validated self-rated 12-item assessment of successful aging and psychological well-being among older adults. Participants will be instructed to select an answer that most closely reflect their attitude towards each statement on a Likert scale from 1 (strongly disagree) to 6 (strongly agree). Scores may range from 6-72, in which a higher score indicates greater life satisfaction.
Shape-Color Sorting | Baseline and 6 months
  The investigators will assess 6-month changes in the Mobile Toolbox "Shape-Color Sorting" test as a measure of cognitive flexibility, a component of executive function (individual cognitive domain). Participants are primary scored on rate correct per second, using the number of correct trials per second as a derived score. Scores may range from 0-10, in which a higher score indicates better cognitive flexibility.
Arrow Matching | Baseline and 6 months
  The investigators will assess 6-month changes in the Mobile Toolbox "Arrow Matching" test as a measure of inhibitory control, a component of executive function (individual cognitive domain). Participants are primary scored on rate correct per second, using the number of correct trials per second as a derived score. Scores may range from 0-10, in which a higher score indicates better inhibitory control.
Faces and Names | Baseline and 6 months
  The investigators will assess 6-month changes in the Mobile Toolbox "Faces and Names" test as a measure of associative memory (individual cognitive domain). The test consists of one encoding phase and three memory phases: Face Recognition, Name Recall, and Name Recognition. A total score is calculated by adding together each component score, for a total of 12 possible points. Scores may range from 0-12, in which a higher score indicates better associative memory.
Body weight | Baseline and 6 months
  The investigators will assess 6-month changes in body weight (in lbs).
Lipid profile | Baseline and 6 months
  The investigators will assess 6-month changes in lipid profiles, including total cholesterol, low-density lipoprotein cholesterol (Friedewald calculated), high-density lipoprotein cholesterol, and triglycerides. All lipids will be reported as mg/dL.
Fasting blood glucose | Baseline and 6 months
  The investigators will assess 6-month changes in fasting blood glucose (in mg/dL).
Insulin-like growth factor-1 | Baseline and 6 months
  The investigators will assess 6-month changes of insulin-like growth factor-1 in the blood (in ng/mL).
Interleukin-6 | Baseline and 6 months
  The investigators will assess 6-month changes of interleukin-6 in the blood (in pg/mL).
Arranging Pictures | Baseline and 6 months
  The investigators will assess 6-month changes in the Mobile Toolbox "Arranging Pictures" test as a measure of episodic memory (individual cognitive domain). This test scores the sum of adjacent pairs correctly placed across two trials. Scores range from 0-26 (14 images results in a maximum of 13 adjacent pairs correct per trial), in which a higher score indicates better episodic memory.
Sequences | Baseline and 6 months
  The investigators will assess 6-month changes in the Mobile Toolbox "Sequences" test as a measure of working memory (individual cognitive domain). This score is the total number of items (individual sequence) correctly answered. The possible score range is 0-30, in which a higher score indicates better working memory.
Number-Symbol Match | Baseline and 6 months
  The investigators will assess 6-month changes in the Mobile Toolbox "Number-Symbol Match" test as a measure of processing speed (individual cognitive domain). The test includes 144 total items, with up to 16 successive screens of 9 items each presented, and examinees have 90 seconds to complete as many items as possible. This score is the total number of items correctly answered in 90 seconds. The possible score range is 0-144, in which a higher score indicates better processing speed.
Waist circumference | Baseline and 6 months
  The investigators will assess 6-month changes in waist circumference (in inches).

OTHER OUTCOMES:
Lutein | Baseline and 6 months
  The investigators will assess 6-month changes in plasma lutein (in µmol/L) as a marker of compliance with pistachio consumption. Participants in the pistachio group are expected to have increases in plasma lutein levels, while participants in the usual group are expected to have no changes.
Gamma tocopherol | Baseline and 6 months
  The investigators will assess 6-month changes in plasma gamma tocopherol (mg/L) as a marker of compliance with pistachio consumption. Participants in the pistachio group are expected to have increases in plasma gamma tocopherol levels, while participants in the usual group are expected to have no changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided